CLINICAL TRIAL: NCT01866267
Title: A Study in HIV+ Patients With CCR5-tropic Virus and Undetectable Viral Load on a First, Non-Selzentry®-Containing Regimen, Switching Them to Once-daily Selzentry® (600mg qd) Plus the Same 2 NRTIs Previously Administered
Brief Title: Switching Undetectables to Selzentry
Acronym: SUDS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Hope Foundation (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUDS_GSK117335
Record Dates: First submitted 2013-02-12; First posted 2013-05-31 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Human Immunodeficiency Virus; AIDS
Keywords: Human Immunodeficiency Virus; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Maraviroc (Other): Patients infected with CCR5 tropic virus that have achieved an undetectable viral load on a non-Selzentry®-containing regimen [Protease Inhibitor (PI)/Non-Nucleoside Reverse Transcriptase Inhibitor (NNRTI)/Integrase Inhibitor plus 2 Nucleoside Reverse Transcriptase Inhibitor (NRTI)] are switched to once-daily Selzentry® (600mg qd) plus the same 2 NRTIs previously administered.
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — HIV positive patients infected with CCR5 tropic virus that have achieved an undetectable viral load on a non-Selzentry®-containing regimen [Protease Inhibitor (PI)/Non-Nucleoside Reverse Transcriptase Inhibitor (NNRTI)/Integrase Inhibitor plus 2 Nucleoside Reverse Transcriptase Inhibitor (NRTI)] are switched to once-daily Selzentry® (600mg qd) plus the same 2 NRTIs previously administered.
  Other Names: Selzentry®; Celsentri®

SUMMARY:
This pilot single arm, single site, open-labeled switch study seeks to enroll thirty (30) HIV positive patients infected with CCR5 tropic virus that have achieved an undetectable viral load on a non-Selzentry®-containing regimen [Protease Inhibitor (PI)/Non-Nucleoside Reverse Transcriptase Inhibitor (NNRTI)/Integrase Inhibitor plus 2 Nucleoside Reverse Transcriptase Inhibitor (NRTI)] and switch them to once-daily Selzentry® (600mg qd) plus the same 2 NRTIs.

DETAILED DESCRIPTION:
The objective of the study is to determine if regimen tolerability/toxicity can be maintained or improved while maintaining virologic suppression following a switch to once-daily Selzentry®.

The study duration is 48 weeks. Patients must have an HIV-1 RNA <100 copies/mL for ≥3 months on their first HIV treatment regimen. Prior regimen modifications for reasons other than virologic failure are acceptable if any previously achieved virologic suppression has been maintained. A Trofile® DNA will be used to document exclusive CCR5 tropism. Patients with history of dual/mixed or CXCR4-tropic HIV-1 are excluded from participation. Patients with prior exposure to Selzentry® are also excluded. Patients that qualify for participation will discontinue the PI, NNRTI, or Integrase inhibitor portion of their regimen and begin Selzentry® 600mg QD. Patients will continue the two (2) NRTIs from the previous treatment regimen.

The primary endpoints is: the percentage of HIV positive patients with undetectable viral load (HIV-1 RNA <100 copies/mL) at Week 24.

Secondary endpoints are: the safety and tolerability of once-daily Selzentry® through Weeks 24 and 48(as measured by clinical and laboratory adverse events and regimen satisfaction questionnaire), the percentage of HIV positive patients with undetectable viral load (HIV-1 RNA < 100 copies/mL) at Week 48, the change from baseline in CD4+ T-cell counts at Weeks 24 and 48, the change from baseline in inflammatory markers (C-reactive protein) at Weeks 24 and 48, and assessment of resistance-associated mutations or viral tropism changes from baseline, if any, emerging at virologic failure.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Are capable of understanding and have signed an informed consent
* Have documented HIV-1 infection by confirmatory laboratory
* Have no acquired immunodeficiency syndrome (AIDS)-defining events in the 3 months before screening, other than cutaneous Kaposi's sarcoma or wasting syndrome due to HIV
* Are able and willing to comply with all protocol requirements and procedures
* Have HIV-1 RNA <100 copies/mL and documented CCR5 tropic virus
* Are receiving their first highly active antiretroviral regimen for at least 12 weeks before screening and are willing to continue that regimen until the baseline visit (previous regimen modifications for reasons other than virologic failure are acceptable if any previously achieved virologic suppression has been maintained)
* Antiretroviral regimen is composed of one NNRTI, one PI (including boosted PIs), or one integrase inhibitor AND two (2) NRTIs

Exclusion Criteria:

* Any history of virologic failure or resistance associated mutations on prior resistance testing
* Any history of dual/mixed- or CXCR4-tropic HIV-1
* Any history of an active AIDS-defining illness per Category C conditions according to the Center for Disease Control (CDC) Classification System for HIV Infection, with the following exceptions: cutaneous Kaposi's sarcoma and wasting syndrome due to HIV
* Any significant diseases (other than HIV-1 infection) or clinically significant findings, including psychiatric and behavioral problems, determined from screening, medical history and/or physical examination that, in the investigator's opinion, would preclude the patient from participating in this study
* Any significant acute illness within 1 week before the initial administration of study drug
* Any active infection secondary to HIV requiring acute therapy; however, patients that require maintenance therapy (i.e. secondary prophylaxis for opportunistic infections) will be eligible for the study
* HCV infection requiring treatment during the study period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Once-Daily Selzentry® through Week 24 | At Week 24
  Percentage of HIV positive patients with Undetectable Viral load (HIV-1 RNA < 100 copies/mL) on once-daily Selzentry plus 2 NRTI

SECONDARY OUTCOMES:
Effectiveness of once-daily Selzentry® through Week 48 | At Week 48
  The percentage of HIV positive patients with undetectable viral load (HIV-1 RNA < 100 copies/mL) on once-daily Selzentry plus 2 NRTI at Week 48
The safety of once-daily Selzentry® through Weeks 24 and 48 | Through Weeks 24 and 48
  The safety of once-daily Selzentry® plus 2 NRTI measured by the frequency and severity of drug-related adverse events (including laboratory abnormalities) through Weeks 24 and 48 of the study.
The change from baseline in CD4+ T-cell counts | at Weeks 24 and 48
  A change from the baseline measurement in CD4+ T-cell counts at Weeks 24 and 48 of the study.
The change from baseline in inflammatory markers (C-reactive protein) | at Weeks 24 and 48
  The change from the baseline measurement in inflammatory markers (C-reactive protein) at Weeks 24 and 48 of the study.
Resistance-Associated Mutations or Tropism Changes from Baseline | at Weeks 24 and 48
  Assessment of any resistance-associated mutations or changes in viral tropism compared to baseline, if any, that emerge upon the occurrence of virologic failure.
Tolerability of Once-Daily Selzentry® | Through Weeks 24 and 48
  The tolerability of once-daily Selzentry® plus 2 NRTI as measured by patient responses to the treatment regimen satisfaction questionnaire, assessed at Weeks 24 and 48 of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley T. Lewis, M.D., MPH, Principal Investigator — St. Hope Foundation, Inc.
Locations (1):
- St. Hope Foundation, Inc., Bellaire, Texas, United States

REFERENCES:
- See also: Health Psychology Research, LTD - source of HIV treatment regimen satisfaction assessment instrument — http://www.healthpsychologyresearch.com